CLINICAL TRIAL: NCT06484595
Title: Guiding Participation Toward Understanding, Inclusion, Diversity, and Equity for Cancer Clinical Trials (GUIDE) Pilot Trial
Brief Title: Clinical Trial Navigation to Increase Participation and Diversity in Cancer Clinical Trials
Acronym: GUIDE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: Andy Hill Cancer Research Endowment (CARE) Fund (Unknown); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: RG1124291; NCI-2024-04530 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P30CA015704 (NIH)
Record Dates: First submitted 2024-06-21; First posted 2024-07-03 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Hematopoietic and Lymphatic System Neoplasm; Malignant Solid Neoplasm
MeSH Terms: interventions — Practice Guidelines as Topic; Standard of Care; Patient Navigation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ARM I (Clinical trial navigator, SOC) (Experimental): Patients meet with a clinical trial navigator to understand activities involved with clinical trials, identify financial barriers to clinical trial participation, and review available financial resources. Patients receive ongoing access to the Guide via a check in meeting once monthly for up to 6 months. Patients also receive SOC supportive care services.
  Interventions: Other: Best Practice; Behavioral: Patient Navigation
- Arm II (SOC) (Active Comparator): Patients receive SOC supportive care services.
  Interventions: Other: Best Practice

INTERVENTIONS:
Other: Best Practice — Receive SOC supportive care services
  Other Names: standard of care; standard therapy
Behavioral: Patient Navigation — Receive clinical trial navigator guide services
  Other Names: Patient Navigator Program
  Arms: ARM I (Clinical trial navigator, SOC)

SUMMARY:
This clinical trial evaluates a clinical trial navigation intervention to help increase participation and diversity in cancer clinical trials. Cancer clinical trials are an important part of the development of treatments, and improved patient care and outcomes. Despite this, only a small number of cancer patients participate in clinical trials. There are many different items that contribute to low clinical trial participation, including health-related social needs (HRSN) and financial burden. Guiding participation toward understanding, inclusion, diversity, and equity for cancer clinical trials (GUIDE), is a program that uses a trained clinical trial navigator, or "Guide", to work with identified potential cancer clinical trial patients to help them recognize and remove HRSN and financial barriers preventing clinical trial participation. A clinical trial navigation intervention, like GUIDE, may help increase participation and diversity in cancer clinical trials.

DETAILED DESCRIPTION:
OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients meet with a clinical trial navigator to understand activities involved with clinical trials, identify financial barriers to clinical trial participation, and review available financial resources. Patients receive ongoing access to the Guide for up to 6 months. Patients also receive standard of care (SOC) supportive care services.

ARM II: Patients receive SOC supportive care services.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years of age
* Identified as potentially eligible for an open clinical trial by clinical trial pre-screening
* Have ≥ 1 health related social need, defined by

  * Food insecurity, housing instability, transportation challenges, or financial instability documented in the Supportive Cancer Care Questionnaire in Epic Electronic Medical Record (EPIC), OR
  * Concerns about insurance, cost of trial, additional trial visits, travel, transportation, childcare/eldercare, OR unable to take time off work, etc., as documented by clinical trial pre-screening (CTPS) or provider, OR
  * Medicaid insurance (including Medicaid pending) documented in EPIC, OR
  * Respond affirmatively (yes, maybe, possibly, I think so, etc.) to the social needs screening question asked by our Research Coordinator: "During your cancer treatment, are you interested in assistance with transportation, food, housing, financial resources, or other barriers to treatment?"
* Able to speak English

Exclusion Criteria:

* Unable to speak English
* Children, adolescents, and teens under the age of 18 years
* Patients participating on clinical trials providing financial navigation, such as clinicaltrials.gov identifier (CT ID): NCT04960787
* Patients refusing to sign Health Insurance Portability and Accountability Act (HIPAA) authorization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2024-09-23 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients in each arm that enroll in a clinical trial | 6 months post-baseline
  Will use descriptive statistics to characterize and compare by pilot trial arm all patients enrolled versus not enrolled in clinical trials. Will be comparing X% of individuals enrolled in a cancer clinical trial (x/50) in the intervention arm and Y% of individuals enrolled in a cancer clinical trial (y/50) in the usual care arm. Information about trial enrollment and retention at 6 months will be abstracted from Online Collaborative Research Environment (OnCore) Clinical Management System.
Proportion of patients in each arm retained to a clinical trial | 6 months post-baseline
  Will use descriptive statistics to characterize and compare by pilot trial arm all patients retained versus not retained in clinical trials. Assessment of trial retention will be restricted to the denominator of patients who enroll in a cancer clinical trial. Information about trial enrollment and retention at 6 months will be abstracted from OnCore Clinical Management System.
Patient trust | 6 months post-baseline
  Will be measured by the 12-item Trust in Medical Researchers scale. Each item will be answered on a 5-point Likert scale and scored accordingly (1 = strongly disagree, 2 = disagree, 3 = neutral, 4 = agree, 5 = strongly agree).
Health related quality of life | 6 months post-baseline
  Will be measured using the Patient Reported Outcomes Measurement Information System (PROMIS) Global Health Score. The PROMIS Global Health instruments generate scores that are converted to T-scores, with a mean of 50 and a standard deviation of 10 in the US general population, allowing for comparison to a reference group. Higher T-scores indicate better health outcomes.
Resilience | 6 months post-baseline
  Will be assessed using the Brief Connor-Davidson Resilience Scale to assess the ability to recover or bounce back from stress.
Resolution of health-related social needs | 6 months post-baseline
  Will be measured by comparing the responses to the Health Related Social Needs (HRSN) questions (food insecurity, housing instability, transportation challenges, financial distress).
Financial burden | 6 months post-baseline
  Will be measured from the patient perspective using the Functional Assessment of Chronic Illness Therapy-Comprehensive Score for financial Toxicity (FACIT-COST) scale. FACIT-COST Includes 12 items with responses on a 5-point Likert type scale. The maximum and minimum total scores range from 0-44 with higher scores representing better financial wellbeing.
Participant perceptions of the intervention (acceptability, appropriateness, feasibility) | At 6 months
  Acceptability, appropriateness, and feasibility of the intervention will be assessed as potential themes in the qualitative interviews with patients in the GUIDE intervention arm of the trial.

SECONDARY OUTCOMES:
Staff time and effort to deliver intervention | At 6 months
  This is the time spent by the Guide with patients, preparing for patient visits, and delivering the intervention.
Participant time costs | At 6 months
  This is the time spent by patients on all activities related to the cancer clinical trial and with the Guide.
Overhead | At 6 months
  Overhead costs are defined as the indirect expenses associated with delivering the GUIDE intervention. This includes the facility costs, measured using the facilities and administration rate, as well as non-clinical equipment and supplies needed to deliver the intervention. Observation-based costs accrued over the intervention delivery period will be averaged and standardized to US 2024 dollars.
Amount of money provided to participants for reimbursement of trial-related expenses | At 6 months
  The amount of money provided to participants for reimbursement of trial-related expenses.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Mendoza, MD, MPH, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2025-05-14): https://cdn.clinicaltrials.gov/large-docs/95/NCT06484595/ICF_000.pdf